CLINICAL TRIAL: NCT00007371
Title: Hepatitis C in Clinically Discordant Hemophilic Siblings
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 954; R01HL064817 (NIH)
Record Dates: First submitted 2000-12-19; First posted 2000-11-28 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2005-01

CONDITIONS: Blood Disease; Hemophilia A; Hepatitis, Viral, Human
MeSH Terms: conditions — Hematologic Diseases; Hemophilia A; Hepatitis, Viral, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
To define the natural history, immunologic, and genetic factors that influence the clinical outcome of hepatitis C in a cohort of hemophilic siblings.

DETAILED DESCRIPTION:
BACKGROUND:

The clinical spectrum of hepatitis C is variable and the factors responsible for these divergent outcomes with chronic hepatitis C infection remain unknown. Dr. Fried and his colleagues are studying a cohort of hemophilic siblings infected with hepatitis C to define the natural history, immunologic, and genetic factors that influence its clinical outcome. Patients with hemophilia have a prevalence rate of hepatitis C as high as 90 percent. The sex-linked pattern of inheritance of hemophilia allows them to identify a cohort of siblings both of who have been infected with hepatitis C. Hemophilic siblings are an attractive population to study because: 1) They are all males; 2) Siblings are relatively close in age; 3) The mode of HCV acquisition is identical; 4) The age at acquisition of hepatitis C is similar 5) The date of acquisition can be confidently estimated upon their factor replacement history; 6) Hemophilic sibs share significant amounts of genetic material.

The study is in response to a Request for Applications entitled "Hepatitis C: Natural History, Pathogenesis, Therapy and Prevention" issued by the National Institute of Diabetes and Digestive and Kidney Diseases

DESIGN NARRATIVE:

Hemophilic siblings with hepatitis C undergo a detailed clinical evaluation to stage their liver disease and to identify sibling pairs with clinically and/or histologically discordant levels of disease activity. These siblings pairs are further studied to define antigen recognition patterns of lymphocyte cells including peripheral CD8 plus cytotoxic T lymphocytes (CTL) and CD4 plus cells and determine their functional significance. Using peripheral blood mononuclear cells, CD8 plus cells are assayed for CTL activity against three overlapping vaccinia/hepatitis C virus (HCV) constructs covering the entire HCV genome followed by fine cloning to identify HCV-specific CTL epitopes. Peripheral CD4 plus cells are tested for their ability to proliferate to HCV antigens. Using stimulation index, Drs. Fried and colleagues are quantitating the presence and magnitude of this response. They are also trying to identify immunodominant regions targeted by cytotoxic T cells using HLA class I matched hemophilic siblings. Finally, they are identifying specific host genes that are preferentially expressed or repressed in patients with delayed progression of their HCV disease. They are quantitating the expression of mRNAs encoding host antiviral defense and immunoregulatory elements in peripheral blood mononuclear cells (PBMCs) and liver tissue from sibling pairs that have discordant chronic hepatitis C using mRNA libraries that are screened by high density oligonucleotide arrays. The expression levels of these genes (including, but not limited to, interferon alpha, beta, and gamma; IRF-1 and IRF-2; interferon induced protein kinase; the cellular protein activator of PKR (PACT) RNase L; interferon-inducible RNA-specific adenosine deaminase; a ribonuclease specific for inosine- containing RNA; chemokine receptors CCR1, CCR3, CCR5, and their signal transduction elements; 2'-5'-oligoadenylate synthetase; tumor necrosis factor; FAS receptor; signal transduction components of these antiviral pathways, and both type 1 and 2 cytokines) are correlated with delayed progression and diminished pathogenesis in paired hemophilic siblings.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fried, Principal Investigator — University of North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kweon YO, Goodman ZD, Dienstag JL, Schiff ER, Brown NA, Burchardt E, Schoonhoven R, Brenner DA, Fried MW. Decreasing fibrogenesis: an immunohistochemical study of paired liver biopsies following lamivudine therapy for chronic hepatitis B. J Hepatol. 2001 Dec;35(6):749-55. doi: 10.1016/s0168-8278(01)00218-5. PMID 11738102
- [Background] Nelson DR, Soldevila-Pico C, Reed A, Abdelmalek MF, Hemming AW, Van der Werf WJ, Howard R, Davis GL. Anti-interleukin-2 receptor therapy in combination with mycophenolate mofetil is associated with more severe hepatitis C recurrence after liver transplantation. Liver Transpl. 2001 Dec;7(12):1064-70. doi: 10.1053/jlts.2001.29414. PMID 11753908
- [Background] Fried MW. Side effects of therapy of hepatitis C and their management. Hepatology. 2002 Nov;36(5 Suppl 1):S237-44. doi: 10.1053/jhep.2002.36810. PMID 12407599
- [Background] Fried MW, Peter J, Hoots K, Gaglio PJ, Talbut D, Davis PC, Key NS, White GC, Lindblad L, Rickles FR, Abshire TC. Hepatitis C in adults and adolescents with hemophilia: a randomized, controlled trial of interferon alfa-2b and ribavirin. Hepatology. 2002 Oct;36(4 Pt 1):967-72. doi: 10.1053/jhep.2002.35529. PMID 12297845
- [Background] Nelson DR, Tu Z, Soldevila-Pico C, Abdelmalek M, Zhu H, Xu YL, Cabrera R, Liu C, Davis GL. Long-term interleukin 10 therapy in chronic hepatitis C patients has a proviral and anti-inflammatory effect. Hepatology. 2003 Oct;38(4):859-68. doi: 10.1053/jhep.2003.50427. PMID 14512873
- [Background] Liu C, Zhu H, Tu Z, Xu YL, Nelson DR. CD8+ T-cell interaction with HCV replicon cells: evidence for both cytokine- and cell-mediated antiviral activity. Hepatology. 2003 Jun;37(6):1335-42. doi: 10.1053/jhep.2003.50207. PMID 12774012
- [Background] Zhu H, Zhao H, Collins CD, Eckenrode SE, Run Q, McIndoe RA, Crawford JM, Nelson DR, She JX, Liu C. Gene expression associated with interferon alfa antiviral activity in an HCV replicon cell line. Hepatology. 2003 May;37(5):1180-8. doi: 10.1053/jhep.2003.50184. PMID 12717400
- [Background] Cabrera R, Tu Z, Xu Y, Firpi RJ, Rosen HR, Liu C, Nelson DR. An immunomodulatory role for CD4(+)CD25(+) regulatory T lymphocytes in hepatitis C virus infection. Hepatology. 2004 Nov;40(5):1062-71. doi: 10.1002/hep.20454. PMID 15486925
- [Background] Theodore D, Fried MW, Kleiner DE, Kroner BL, Goedert JJ, Eyster ME, Faust SP, Sherman KE, Kessler CM, Francis C, Aledort LM. Liver biopsy in patients with inherited disorders of coagulation and chronic hepatitis C. Haemophilia. 2004 Sep;10(5):413-21. doi: 10.1111/j.1365-2516.2004.00919.x. PMID 15357765